CLINICAL TRIAL: NCT02569450
Title: The Impact of Surgical Outcomes Monitoring Using Control Chart on Surgical Performance: A Cluster Randomized Trial
Brief Title: Evaluation of Control Chart Impact on Surgical Outcomes
Acronym: SHEWHART
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0282
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Digestive Surgery
Keywords: Surgery; Performance; Outcome; Control chart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention arm: Hospitals randomly assigned to the intervention arm with surgical outcomes monitoring
  Interventions: Behavioral: Surgical outcomes monitoring using Shewhart control chart
- Hospitals in control arm: Hospitals randomly assigned to the control arm without surgical outcome monitoring

INTERVENTIONS:
Behavioral: Surgical outcomes monitoring using Shewhart control chart — * Assistance by a local surgeon responsible for the implementation of intervention within his/her department
  * Quarterly team meeting to interpret variations in observed outcomes on the control charts
  * Restitution of surgical outcomes based on wall posters in operating room
  * Training sessions provided to local surgeon for appropriate control chart utilization
  Groups: Intervention arm

SUMMARY:
This two arms parallel cluster-randomized trial will evaluate the impact of monitoring surgical outcomes using Shewhart control chart (intervention) on the occurence of major adverse events, among a large sample of French surgical departments. Trends in surgical outcomes before and after the intervention will be compared between arms.

ELIGIBILITY:
Inclusion Criteria:

- All adults needing a digestive surgery who are hospitalized in one of the 40 departments

Exclusion Criteria:

* Age < 18 years old
* Hospitalization <24 hours
* Absence of surgical procedure
* Ambulatory care
* Palliative care
* Organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients operated in participating French public and private hospitals (cluster)
Sampling Method: Non-Probability Sample
Enrollment: 157594 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of any major adverse event during hospitalization | within 30 days following surgical procedure
  Major adverse events include postoperative death, complication, unplanned intensive care stay or reoperation within 30 days of surgery.

SECONDARY OUTCOMES:
Occurrence of any death during hospitalization within 30 days of surgery | within 30 days following surgical procedure
Occurrence of any complication during hospitalization within 30 days of surgery | at the end of hospitalization
Occurrence of unplanned intensive care stay during hospitalization within 30 days of surgery | within 30 days following surgical procedure
Occurrence of reoperation during hospitalization within 30 days of surgery | within 30 days following surgical procedure
Number of hospital bed-days consumed | within 30 days following surgical procedure
Hospitalization costs from a health insurance perspective | within 30 days following surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Pôle IMER, Lyon, France

REFERENCES:
- [Derived] Skinner S, Pascal L, Polazzi S, Chollet F, Lifante JC, Duclos A; SHEWHART Trial Group. Economic analysis of surgical outcome monitoring using control charts: the SHEWHART cluster randomised trial. BMJ Qual Saf. 2024 Apr 24;33(5):284-292. doi: 10.1136/bmjqs-2022-015390. PMID 37553238
- [Derived] Duclos A, Chollet F, Pascal L, Ormando H, Carty MJ, Polazzi S, Lifante JC; SHEWHART Trial Group. Effect of monitoring surgical outcomes using control charts to reduce major adverse events in patients: cluster randomised trial. BMJ. 2020 Nov 4;371:m3840. doi: 10.1136/bmj.m3840. PMID 33148601